CLINICAL TRIAL: NCT04189276
Title: A Phase II Clinical Trial to Evaluate the Safety and Efficacy of Therapeutic Hepatitis B Adenovirus Injection (T101) Combined With Nucleoside (Acid) Analogues in Chronic Hepatitis B Patients
Brief Title: Safety and Efficacy of Therapeutic Hepatitis B Adenovirus Injection (T101) Combined With Nucleoside (Acid) Analogues in Chronic Hepatitis B Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tasly Tianjin Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSL-BM-T101-II
Record Dates: First submitted 2019-11-03; First posted 2019-12-06 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Hepatitis B Virus (HBV)
Keywords: Hepatitis B Virus (HBV) infection
MeSH Terms: conditions — Hepatitis B; Infections | interventions — entecavir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group1 (Active Comparator): T101+ETV(Entecavir) /TDF(Tenofovir)
  Interventions: Biological: ETV/TDF+T101 No.1
- Group2 (Active Comparator): T101+ETV/TDF
  Interventions: Biological: ETV/TDF+T101 No.2
- Group3 (Active Comparator): ETV or TDF
  Interventions: Biological: ETV or TDF
- Group4 (Active Comparator): Peg-IFNα-2b+ETV/TDF
  Interventions: Biological: ETV/TDF+Peg-IFNα-2b

INTERVENTIONS:
Biological: ETV/TDF+T101 No.1 — Patients will be injected with T101 once on Day1 (Week0), Day8 (Week1), Day15 (Week2), Day106 (Week15), Day113 (Week16), Day120 (Week17), Day211 (Week30), Day218 (Week31), Day225 (Week32), Day316 (Week45), Day323 (Week46), Day330 (Week47); ETV or TDF will be administrated once each day successively until Day420.
  Arms: Group1
Biological: ETV/TDF+T101 No.2 — Patients will be injected with T101 once on Day1 (Week0), Day106 (Week15), Day211 (Week30), Day316 (Week45); ETV or TDF will be administrated once each day successively until Day420.
  Arms: Group2
Biological: ETV or TDF — Patients will be administrated ETV or TDF once each day successively until Day420.
  Arms: Group3
Biological: ETV/TDF+Peg-IFNα-2b — Patients will be administrated Peg-IFNα-2b successively once a week until Day330 (Week47); ETV or TDF will be administrated once each day successively until Day420.
  Arms: Group4

SUMMARY:
A multi-center, randomized, open-label, group controlled study to evaluate the safety and efficacy of T101 combined with nucleoside (acid) analogues in chronic hepatitis B patients.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following inclusion criteria to be enrolled in this study:

* 1. Patients between the ages of 18 and 60 years, male or female;
* 2. Body weight is no less than 45kg for female and no less than 50kg for male;
* 3. Meets the diagnosis and treatment standards of chronic hepatitis B in China's 2015 Guidelines for the Prevention and Treatment of Chronic Hepatitis B;
* 4. Currently, should have taken nucleoside (acid) analogues for 1 year or more;
* 5. HBV DNA<100 IU/ml; HBsAg is positive and no more than 3000 IU/ml；HBeAg is negative；
* 6. Be able to understand and sign informed consent.

Exclusion Criteria:

Patients with any of the following items will not be enrolled in this study:

* 1. Pregnant or lactating women; male or female who have planned to have children from the start of the study to sixth month after the end of the study.
* 2. Have received interferon treatment within 6 months prior to the screening;
* 3. Have taken strong immunomodulators (such as adrenocortical hormone, thymosin alpha 1, thymosin 5, etc.) within 6 months before the screening, and the course of treatment was more than 2 weeks;
* 4. Have taken hepatotoxic drugs (such as dapsone, erythromycin, fluconazole, ketoconazole, rifampicin) within 6 months before screening, and the course of treatment was more than 2 weeks;
* 5. Currently or previously diagnosed or suspected with cirrhosis or liver cancer; or AFP > 50ng/ml;
* 6. Liver diseases caused by other causes: including alcoholic hepatitis, drug hepatitis, autoimmune liver disease;
* 7. Currently be infected of HAV, HCV, HDV, HEV, HIV and syphilis;
* 8. Have mental diseases, including but not limited to depression, anxiety, mania, schizophrenia;
* 9. Uncontrolled epilepsy;
* 10. Complicated with serious systemic diseases, including but not limited to: autoimmune diseases (such as psoriasis, systemic lupus erythematosus, etc.); not well controlled cardiovascular disease (such as high blood pressure, unstable angina pectoris, heart failure, etc.), endocrine system disease (such as thyroid function hyperfunction or loss, diabetes, etc.), respiratory system diseases (such as pulmonary infection, chronic obstructive pulmonary disease and pulmonary interstitial diseases, etc.), digestive system diseases (e.g., chronic colitis, etc.), kidney disease (such as chronic kidney disease, renal insufficiency, etc.), blood system diseases (such as autoimmune anemia, hemophilia, etc.); currently or previously diagnosed or suspected with malignant tumor;
* 11. Fundus diseases, such as not well controlled retinopathy, etc.;
* 12. Laboratory neutrophil count<1.5×109/L; platelet count <90×109/L;
* 13. Prothrombin time was extended by more than 3 seconds compared with the upper limit of normal reference value (ULN);
* 14. ALT>1.5×ULN; TBIL>2×ULN; SCR>1.5×ULN; serum creatine kinase >3×ULN; ALB<35g/L;
* 15. ANA>1:1000, anti-smooth muscle antibody>1:1000, thyrotropic hormone receptor antibody >2×ULN;
* 16. Allergic constitution or allergic to experimental drugs and excipients;
* 17. Plan to receive or have already had an organ transplant;
* 18. Participated in any clinical trial or taken any IMP (investigational medical product) within 3 months prior to the trial;
* 19. Other cases that could not be enrolled in the judgement of the investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
All the observed or reported AEs (adverse events) | through study completion, an average of 60 weeks
  observe and record all the AEs of patients during the clinical trial and determine their correlation with the investigational medical product
HBsAg change | Day106 (Week15), Day211 (Week30), Day316 (Week45), Day337 (Week48), Day421 (Week60) after administration
  evaluate the HBsAg change from the baseline to evaluate the efficacy of T101

SECONDARY OUTCOMES:
The percentage of Subjects' HBsAg decrease ≥ 1 log | Day106 (Week15), Day211 (Week30), Day316 (Week45), Day337 (Week48), Day421 (Week60) after administration
  to evaluate the efficacy of T101
The percentage of Subjects' HBsAg decrease ≥ 0.5 log | Day106 (Week15), Day211 (Week30), Day316 (Week45), Day337 (Week48), Day421 (Week60) after administration
  to evaluate the efficacy of T101
Negative convention rate of HBsAg | Day316 (Week45), Day337 (Week48), Day421 (Week60) after administration
  to evaluate the efficacy of T101
Positive convention rate of HBsAb | Day316 (Week45), Day337 (Week48), Day421 (Week60) after administration
  to evaluate the efficacy of T101

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Youan Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Ditan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Tianjin Second People's Hospital, Tianjin, Tianjin Municipality